CLINICAL TRIAL: NCT01534494
Title: Effects and Therapeutic Potential of Psilocybin in Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Heffter Research Institute (Other)
Responsible Party: Principal Investigator, Michael Bogenschutz, Professor of Psychiatry, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Heffter-UNM-HSC-15671
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; psilocybin; clinical trial; motivational enhancement therapy
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- psilocybin (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — two doses of 0.3 mg/kg PO and 0.4 mg/kg PO, separated by 4 weeks in combination with 12 weeks of manualized outpatient psychosocial treatment including preparation, debriefing, and motivational enhancement therapy.

SUMMARY:
This trial is an open-label pilot study (N = 10) designed to assess the effects of psilocybin in alcohol dependent participants, demonstrate the feasibility of the integrated behavioral/pharmacologic intervention, and provide preliminary outcome and safety data. Participants will receive psilocybin orally in two all-day administration sessions, conducted in a secure outpatient psychiatric setting, in a dose range that has been well-tolerated in recent studies. Psilocybin administration will occur in the context of a behavioral intervention including a total of 12 sessions over 12 weeks, incorporating Motivational Enhancement Therapy (MET (Miller, Zweben et al. 1992; Miller 1995), based on Motivational Interviewing (Miller and Rollnick 2002)) with booster sessions, as well as preparation before and debriefing after the psilocybin administration sessions. The MET will incorporate attention to spirituality as well as drinking behavior as a primary subject of change. Drinking outcomes and changes in several potential mediators of treatment effect, including motivation, self-efficacy, craving, depression, anxiety, and spiritual dimensions of the experience, will be measured during treatment and for 24 weeks after the end of treatment. The investigators hypothesize that drinking will decrease following the psilocybin sessions, and that increases in motivation, self-efficacy, and spirituality (primary contrast 12 weeks vs. baseline) will be observed among study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 25-65 with diagnosis of alcohol dependence, as ascertained using the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV version);
2. Concerned about their drinking, but not planning to pursue any other form of treatment at present (12-step meetings are not considered treatment);
3. Able to provide voluntary informed consent;
4. Having at least 2 heavy drinking days in the past 30 days;
5. Willing to commit to the goal of abstinence at least from the time of the first psilocybin administration session until the end of treatment.
6. At least 24 hours abstinence from alcohol at the time of the psilocybin administration sessions;
7. If female of childbearing potential, willing to use approved form of contraception from screening until after the psilocybin administration sessions;
8. Having a family member or friend who can pick them up and stay with them overnight after the psilocybin administration sessions; and
9. Able to provide adequate locator information.

Exclusion Criteria:

1. Exclusionary medical conditions (e.g., seizure disorder, significantly impaired liver function, coronary artery disease, uncontrolled hypertension, history of cerebrovascular accident, severe obesity (BMI greater than or equal to 35);
2. Exclusionary psychiatric conditions (schizophrenia, schizoaffective disorder, bipolar disorder, current major depression, current post-traumatic stress disorder, current suicidality);
3. A family history of schizophrenia, schizoaffective disorder, bipolar disorder, or suicide (first or second degree relatives);
4. Lifetime history of hallucinogen use on more than 10 occasions, or any use in the past 30 days;
5. Cocaine, psychostimulant, or opioid dependence (past 12 months) or current (past 30 days) use;
6. A history of medically significant suicide attempt or violent crime;
7. Significant alcohol withdrawal (CIWA-Ar score greater than 7);
8. Exclusionary laboratory abnormalities (any liver function test (LFT) greater than 5 times normal, ECG evidence of ischemia, serious abnormalities of complete blood count or chemistries);
9. Active legal problems with the potential to result in incarceration;
10. Pregnancy or lactation;
11. The need to take excluded medication (e.g., antidepressants, antipsychotics, psychostimulants, pharmacologic treatments for addictions).
12. High risk of adverse emotional reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, serious current stressors, lack of meaningful social support).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Bogenschutz, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psilocybin
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Psilocybin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 10
Percent Heavy Drinking Days at Screening [Mean (Standard Deviation); unit: Percentage] — Based on 84-day Timeline Followback interview conducted at screening
  Percentage | 35.0006 (19.55541)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Heavy Drinking Days
Time Frame: weeks 5-12 post initiation of treatment vs. 12 weeks prior to treatment
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin
Number analyzed (Participants) | 9
percentage of days | -25.962 (22.398)
Statistical Analysis 1: Comparison: Psilocybin; Single-group pre-post contrast; Test type: Other — Paired t-test; p = 0.008, t-test, 2 sided; Paired t-test for significance of change. t(8) = 3.477. P(2-sided) = 0.008

ADVERSE EVENTS:
Time Frame: 32 weeks following first dose of psilocybin
Groups:
- Psilocybin: This was a single-arm study. All participants were assigned to receive the same schedule of psychotherapy and psilocybin administration, as described in the Protocol section. Arms/Groups cannot be provided for each dose level separately because information was not collected.
Arm/Group | Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (3)

LIMITATIONS AND CAVEATS:
Open-label single-group study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No